CLINICAL TRIAL: NCT01126125
Title: Iodized Oil Supplementation During Infancy
Brief Title: Study of the Effect of Iodized Oil Supplementation During Infancy
Acronym: INSIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SwissFIT
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Iodine Deficiency
Keywords: iodine; infant; breastfeeding; deficiency
MeSH Terms: conditions — Breast Feeding | interventions — Iodized Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodized oil to mother (Experimental): 400 mg iodine as iodized oil to breastfeeding mother
  Interventions: Dietary Supplement: Iodized oil
- Iodized oil to infant (Active Comparator): 100 mg of iodine as iodized oil to infant
  Interventions: Dietary Supplement: Iodized oil

INTERVENTIONS:
Dietary Supplement: Iodized oil — 400 mg of iodine vs 100 mg of iodine as iodized oil

SUMMARY:
In iodine-deficient countries or regions that have inadequate iodized salt distribution, the World Health Organization (WHO) recommends choosing one of two methods to improve iodine intakes in breastfeeding infants: 1) iodine supplement (400 mg as iodized oil; 1/year) to the breastfeeding mother, or 2) iodine supplement (100 mg as iodized oil; 1/year) directly to the infant. However, the relative efficacy of these two methods of providing iodine to the newborn has never been directly compared. Whether the first method of iodine supplementation to the breast feeding mother can significantly improve iodine supply and maintain normal thyroid function in her infant remains unclear. This study will directly compare these two strategies. The hypothesis is that the two strategies will be equally effective in providing iodine to the newborn.

DETAILED DESCRIPTION:
In iodine-deficient countries or regions that have inadequate iodized salt distribution, WHO recommends choosing one of two methods to improve iodine intakes in breastfeeding infants:

Method 1) iodine supplement (400 mg as iodized oil; 1/year) to the breastfeeding mother Method 2) iodine supplement (100 mg as iodized oil; 1/year) directly to the infant

However, the relative efficacy of these two methods of providing iodine to the newborn has never been directly compared. Whether the first method of iodine supplementation to the breast feeding mother can significantly improve iodine supply and maintain normal thyroid function in her infant remains unclear.

The mountains of southern Morocco are areas of iodine deficiency. Although the government has been promoting iodization of salt, there are hundreds of small salt producers in the mountains who do not have the funding or infrastructure to iodize their salt, and thus many rural populations still are consuming non-iodized locally-produced salt. At the study site, a 2009 pilot survey of urinary iodine has found that the population in this region is moderately iodine sufficient.

Thus, according to WHO, breastfeeding women and/or their infants should be provided with oral iodine supplementation. But which of the above supplementation methods is preferable? Controlled studies clearly demonstrate that iodine repletion in moderate-to severely iodine deficient school-age children increases insulin-like growth factor (IGF)-1 and insulin-like growth factor binding protein (IGFBP)-3 concentrations and improves somatic growth (height and weight). But whether supplying adequate iodine to iodine deficient infants improves their somatic growth has not been tested.

Therefore, the study hypotheses are: In Moroccan infants who are breastfeeding, method 2 will be more efficacious than method 1 in:

1. increasing urinary iodine (UI) concentrations
2. improving thyroid function (TSH, TT4)
3. increasing IGF-1, IGFBP-3
4. improving somatic growth (length, weight, head circumference)

The study design will be a double-blind, randomized controlled intervention trial in southern Morocco lasting 1 year. Healthy mother-infant pairs (n=240) who are breastfeeding will be recruited while the infant is >1 mo of age. They will be divided into two groups as follows:

1) method 1: mother receives 400 mg of iodine as oral iodized oil + infant receives placebo capsule; or 2) method 2: mother receives placebo capsule + infant receives 100 mg oral iodized oil.

The outcomes will be:

1. length, weight, head circumference
2. IGF-1, IGFBP-3, thyroid functions (TSH, total T4) from a dried blood spot taken from a finger prick in the mothers/heel prick in the infants
3. urinary and breast milk iodine concentrations These samples (blood spot, urine, breastmilk, anthropometry) will be collected during the first year visits of the infant to the local health clinic for routine pediatric vaccinations (at 1, 12, 20 and 40-52 wks).

ELIGIBILITY:
Inclusion Criteria:

* breastfeeding term infant

Exclusion Criteria:

* not breastfeeding
* major medical illnesses

Ages: 4 Weeks to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 241 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Infant height and weight | 1st year after birth

SECONDARY OUTCOMES:
Infant head circumference | 1st year after birth
Thyroid hormone concentrations | 1st year after birth
Urinary iodine concentrations | 1st year after birth
Infant development score | 1st year after birth

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, MD, Principal Investigator — Swiss Federal Institute of Technology Zurich
Locations (1):
- Semilila Faculty of Sciences, Marrakesh, Marrakech, Morocco

REFERENCES:
- [Derived] Bouhouch RR, Bouhouch S, Cherkaoui M, Aboussad A, Stinca S, Haldimann M, Andersson M, Zimmermann MB. Direct iodine supplementation of infants versus supplementation of their breastfeeding mothers: a double-blind, randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2014 Mar;2(3):197-209. doi: 10.1016/S2213-8587(13)70155-4. Epub 2013 Nov 22. PMID 24622750